CLINICAL TRIAL: NCT02651493
Title: Down Syndrome Detection From Facial Photographs Using Machine Learning Techniques
Brief Title: Digital Dysmorphology Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kevin Cleary (Other)
Collaborators: Children's National Research Institute (Other); George Washington University (Other); Chiang Mai University (Other)
Responsible Party: Sponsor-Investigator, Kevin Cleary, PhD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00003506.
Record Dates: First submitted 2015-10-22; First posted 2016-01-11 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — Moire Topography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Down syndrome (Active Comparator): photographs of individuals less than 18 yo with Down syndrome
  Interventions: Device: photographs
- Control group (Active Comparator): photographs of individuals less than 18 yo with a genetic referral (not Down syndrome) or a healthy sibling to a child with Down syndrome
  Interventions: Device: photographs

INTERVENTIONS:
Device: photographs — computer based program to analyze photographs (computer-aided diagnosis (CAD) software)

SUMMARY:
In this study, the investigators propose a novel method to detect Down syndrome using photography for facial dysmorphology, a tool called computer-aided diagnosis (CAD). After validating the method, this technology will be expanded to perform similar functions to assist in the detection of other dysmorphic syndromes.

By using photography and image analysis this automated assessment tool would have the potential to improve the diagnosis rate and allow for remote, non-invasive diagnostic evaluation for dysmorphologists in a timely manner.

DETAILED DESCRIPTION:
In this study, investigators propose a novel method to detect Down syndrome using photography for facial dysmorphology, a tool called computer-aided diagnosis (CAD) . Local texture features based on Contourlet transform and local binary pattern are investigated to represent the facial characteristics. A support vector machine classifier is then used to discriminate between normal and abnormal cases. Accuracy, precision and recall are used to evaluate the method. After validating the method, this technology will then be expanded to perform similar functions to assist in the detection of other dysmorphic syndromes.

By using photography and image analysis this automated assessment tool would have the potential to improve the diagnosis rate and allow for remote, non-invasive diagnostic evaluation for dysmorphologists in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subject with Down syndrome.
* Healthy pediatric siblings of a subject with Down syndrome and/or other individuals with another genetic referral to serve as a control group.
* Subject must be less than 18 years old.

Exclusion Criteria:

* Subjects 18 years or older.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 750 (Estimated)
Dates: Start 2013-02; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Down syndrome accurately assessed by computer-aided detection (CADe) tool | 5 years
  The study will enroll and analyze photographic data from syndromic and non-syndromic cases to investigate the parameters required to achieve an accuracy of the computer-aided detection (CADe) tool for children with genetic syndromes at a level of 90% accuracy.
Number of participants with Down syndrome accurately assessed by computer-aided detection (CADe) tool | 5 years
  The study will enroll and analyze photographic data from syndromic and non-syndromic cases to investigate the parameters required to achieve an accuracy of the computer-aided detection (CADe) tool for children with genetic syndromes at a level of 95% accuracy.

SECONDARY OUTCOMES:
Number of participants with other dysmorphic syndromes accurately assessed by computer-aided detection (CADe) tool | 5 years
  The study will enroll and analyze photographic data from syndromic and non-syndromic cases to investigate the parameters required to achieve an accuracy of the computer-aided detection (CADe) tool for children with genetic syndromes at a level of 90% accuracy.
Number of participants with other dysmorphic syndromes accurately assessed by computer-aided detection (CADe) tool | 5 years
  The study will enroll and analyze photographic data from syndromic and non-syndromic cases to investigate the parameters required to achieve an accuracy of the computer-aided detection (CADe) tool for children with genetic syndromes at a level of 95% accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Cleary, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National, Washington D.C., District of Columbia, United States